CLINICAL TRIAL: NCT01283594
Title: A Double-blind, Randomized, Placebo-controlled Study of the Safety and Efficacy of SYN115 as Adjunctive Therapy in Levodopa-treated Parkinson's Subjects With End of Dose Wearing Off
Brief Title: Safety and Efficacy Study of SYN115 in Parkinson's Patients Using Levodopa to Treat End of Dose Wearing Off
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biotie Therapies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYN115-CL02
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2014-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — tozadenant; BID protein, human; Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Tozadenant (SYN115) 60 mg BID (Experimental): Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Interventions: Drug: Tozadenant (SYN115) 60 mg BID; Drug: Levodopa (L-dopa)
- Tozadenant (SYN115) 120 mg BID (Experimental): Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Interventions: Drug: Levodopa (L-dopa); Drug: Tozadenant (SYN115) 120 mg BID
- Tozadenant (SYN115) 180 mg BID (Experimental): Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Interventions: Drug: Levodopa (L-dopa); Drug: Tozadenant (SYN115) 180 mg BID
- Tozadenant (SYN115) 240 mg BID (Experimental): Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Interventions: Drug: Levodopa (L-dopa); Drug: Tozadenant (SYN115) 240 mg BID
- Sugar Pill (Placebo Comparator): White-coated, modified-oval placebo tablets.
  Interventions: Drug: Placebo; Drug: Levodopa (L-dopa)

INTERVENTIONS:
Drug: Tozadenant (SYN115) 60 mg BID — Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Total daily doses include 60 mg BID.
  Arms: Tozadenant (SYN115) 60 mg BID
Drug: Placebo — White-coated, modified-oval placebo tablets.
  Arms: Sugar Pill
Drug: Levodopa (L-dopa) — One intravenous infusion of L-dopa to reach approximately 600 ng/ ml plasma concentration.
  Other Names: L-dopa
Drug: Tozadenant (SYN115) 120 mg BID — Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Total daily doses include 120 mg BID.
  Arms: Tozadenant (SYN115) 120 mg BID
Drug: Tozadenant (SYN115) 180 mg BID — Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Total daily doses include 180 mg BID.
  Arms: Tozadenant (SYN115) 180 mg BID
Drug: Tozadenant (SYN115) 240 mg BID — Tozadenant tablets, white-coated, modified-oval tablets manufactured in 60 mg dosage strengths.
  Total daily doses include 240 mg BID.
  Arms: Tozadenant (SYN115) 240 mg BID

SUMMARY:
The purpose of this research study is to test the effect of SYN115 compared to placebo (a "sugar pill" that looks like SYN115 but does not include active drug) on movement during the "on" and "off" states as well as other symptoms that some patients with Parkinson's disease experience. This study will also look at whether or not patients with Parkinson's disease experience "side-effects" with SYN115.

ELIGIBILITY:
Inclusion Criteria:

* Meet Parkinson's Disease (PD) diagnosis consistent with UK PD diagnostic criteria
* Meet Hoehn and Yahr PD stage
* Good response to levodopa
* Stable regimen of anti-parkinson medications
* Are able to complete a Parkinson's disease diary
* If of childbearing potential(male and female), use an acceptable method of birth control
* Able and willing to sign an IRB/IEC approved informed consent
* Able and willing to understand study requirements, follow study instructions, attend all visits and undergo all planned tests.

Exclusion Criteria:

* Secondary or atypical Parkinson's
* Neurosurgical intervention for Parkinson's disease
* Treatment with apomorphine
* Treatment with anti-psychotic drugs
* Other abnormal findings on physical or neuro exam or history that in the opinion of the investigator would make subject unsuitable for the study or prejudice safety and efficacy evaluation
* MMSE less than 26
* Subjects with untreated or uncontrolled current episode of major depression
* Receipt of any anti-psychotic drugs greater than 1 month in the past 5 years or any exposure in past year (except for quetiapine at doses <100mg per day)
* Women pregnant or lactating
* History of hepatitis, cholangitis
* Untreated or uncontrolled hypothyroidism or hyperthyroidism
* Drops in blood pressure requiring medication to maintain blood pressure
* Any clinically significant out of range laboratory evaluations
* Known sensitivity to the study medication or its components
* Suicide ideation or type 4 or type 5 on the Columbia suicide severity rating scale
* Finding of malignant melanoma on full body skin exam
* Impulse disorder conditions

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Assess efficacy of different doses of SYN115 for reducing the mean total hours of awake time per day spent in the off state | 12 weeks

SECONDARY OUTCOMES:
To assess the effect of SYN115 on dyskinesia | 12 weeks
To assess the effect of SYN115 on UPDRS scores | 12 weeks
To assess investigator and patient impressions of PD severity and change | 12 weeks
To assess the effect of SYN115 on non motor symptoms of PD | 12 weeks
To assess the safety and tolerability of SYN115 | 12 weeks
To assess the effects of SYN115 on daytime drowsiness, impulsive behavior, development of melanoma and suicidal ideation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steve Bandak, MD, Study Chair — Biotie Therapies Inc.; Ann Neale, RN, Study Director — Biotie Therapies Inc.
Locations (61):
- United States (40):
  - Birmingham, Alabama
  - La Jolla, California
  - Loma Linda, California
  - Los Angeles, California
  - Oxnard, California
  - San Francisco, California
  - Denver, Colorado
  - Manchester, Connecticut
  - New Haven, Connecticut
  - Boca Raton, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Boise, Idaho
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - West Bloomfield, Michigan
  - Minneapolis, Minnesota
  - Commack, New York
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Roanoke, Virginia
  - Milwaukee, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Santa Fe
- Canada (5):
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - Ottawa, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Chile (2):
  - Santiago
  - Valdivia
- Romania (5):
  - Brasov
  - Bucharest
  - Constanța
  - Târgu Mureş
  - Timișoara
- Ukraine (7):
  - Dnipropetrovsk
  - Donetsk
  - Kiev
  - Lviv
  - Poltava
  - Vinnytsia
  - Zaporizhzhya

REFERENCES:
- [Derived] Hauser RA, Olanow CW, Kieburtz KD, Pourcher E, Docu-Axelerad A, Lew M, Kozyolkin O, Neale A, Resburg C, Meya U, Kenney C, Bandak S. Tozadenant (SYN115) in patients with Parkinson's disease who have motor fluctuations on levodopa: a phase 2b, double-blind, randomised trial. Lancet Neurol. 2014 Aug;13(8):767-76. doi: 10.1016/S1474-4422(14)70148-6. Epub 2014 Jul 6. PMID 25008546